CLINICAL TRIAL: NCT00337194
Title: A Randomized Double-Blinded Placebo Controlled Phase II Study of the Anti-CD30 Antibody, SGN-30 (NSC #731636), in Combination With Gemcitabine, Vinorelbine, and Pegylated Liposomal Doxorubicin (GVD) for Patients With Relapsed/Refractory Hodgkin Lymphoma
Brief Title: SGN-30 and Combination Chemotherapy in Treating Patients With Relapsed or Refractory Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02822; NCI-2012-02822 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CALGB-50502 (Other: Cancer and Leukemia Group B); CALGB-50502 (Other: CTEP); U10CA031946 (NIH); P30CA014236 (NIH)
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2014-10

CONDITIONS: Adult Lymphocyte Depletion Hodgkin Lymphoma; Adult Lymphocyte Predominant Hodgkin Lymphoma; Adult Mixed Cellularity Hodgkin Lymphoma; Adult Nodular Sclerosis Hodgkin Lymphoma; Recurrent Adult Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — SGN-30 monoclonal antibody; Brentuximab Vedotin; Vinorelbine; liposomal doxorubicin; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Arm I (SGN-30, chemotherapy) (Experimental): Participants receive one of the following regimens every cycle depending on history of prior stem cell transplant. Cycle is 21 days.
  No prior stem cell transplant:
  SGN-30: 12 mg/kg IV days 1 & 8, vinorelbine: 20 mg/m^2 IV days 1 & 8, gemcitabine: 1000 mg/m^2 IV days 1 & 8, pegylated doxorubicin HCl liposome: 15 mg IV days 1 & 8.
  Prior stem cell transplant SGN-30: 12 mg/kg IV days 1 & 8, vinorelbine: 15 mg/m^2 IV days 1 & 8, gemcitabine: 800 mg/m^2 IV days 1 & 8, pegylated doxorubicin HCl liposome: 10 mg IV days 1 & 8.
  Interventions: Biological: monoclonal antibody SGN-30; Drug: vinorelbine tartrate; Drug: pegylated liposomal doxorubicin hydrochloride; Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis; Other: pharmacological study
- Arm II (placebo, chemotherapy) (Active Comparator): Participants receive one of the following regimens every cycle depending on history of prior stem cell transplant. Cycle is 21 days.
  No prior stem cell transplant:
  SGN-30: 12 mg/kg IV days 1 & 8, vinorelbine: 20 mg/m^2 IV days 1 & 8, gemcitabine: 1000 mg/m^2 IV days 1 & 8, pegylated doxorubicin HCl liposome: 15 mg IV days 1 & 8.
  Prior stem cell transplant SGN-30: 12 mg/kg IV days 1 & 8, vinorelbine: 15 mg/m^2 IV days 1 & 8, gemcitabine: 800 mg/m^2 IV days 1 & 8, pegylated doxorubicin HCl liposome: 10 mg IV days 1 & 8.
  Interventions: Other: placebo; Drug: vinorelbine tartrate; Drug: pegylated liposomal doxorubicin hydrochloride; Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: monoclonal antibody SGN-30 — Given IV
  Other Names: SGN-30
  Arms: Arm I (SGN-30, chemotherapy)
Other: placebo — Given IV
  Other Names: PLCB
  Arms: Arm II (placebo, chemotherapy)
Drug: vinorelbine tartrate — Given IV
  Other Names: Eunades; navelbine ditartrate; NVB; VNB
Drug: pegylated liposomal doxorubicin hydrochloride — Given IV
  Other Names: CAELYX; Dox-SL; DOXIL; doxorubicin hydrochloride liposome; LipoDox
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This randomized phase II trial studies the side effects and how well giving monoclonal antibody SGN-30 together with combination chemotherapy works in treating patients with Hodgkin lymphoma that has returned after a period of improvement or did not respond to previous treatment. Monoclonal antibodies, such as SGN-30, may interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as gemcitabine hydrochloride, vinorelbine tartrate, and pegylated liposomal doxorubicin hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving monoclonal antibody SGN-30 together with combination chemotherapy may kill more cancer cells and shrink tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the complete and partial response rates following treatment with the anti-cluster of differentiation (CD) 30 antibody, SGN-30 (monoclonal antibody SGN-30), and gemcitabine (gemcitabine hydrochloride), vinorelbine (vinorelbine tartrate), and pegylated liposomal doxorubicin (pegylated liposomal doxorubicin hydrochloride) (GVD) in patients with relapsed or refractory Hodgkin lymphoma (HL).

II. To assess time to progression and overall survival in patients treated with SGN-30 and GVD in patients with relapsed or refractory Hodgkin lymphoma (HL).

III. To evaluate the toxicity of SGN-30 in combination with GVD in patients with relapsed and refractory HL.

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetic profile of SGN-30 when combined with GVD chemotherapy.

II. To correlate soluble (s) CD30 levels with response to treatment. III. To determine the incidence of human anti-chimeric antibodies (HACA) formation following repetitive SGN-30 dosing.

IV. To correlate Fc gamma receptor polymorphisms with response to treatment.

OUTLINE:

Part 1 (closed to accrual as of 5/18/2007): Patients receive monoclonal antibody SGN-30 intravenously (IV) over 2 hours, vinorelbine tartrate IV over 6-10 minutes, gemcitabine hydrochloride IV over 30 minutes, and pegylated doxorubicin hydrochloride liposome IV over 90 minutes on days 1 and 8. Treatment repeats every 21 days until 10 out of 16 patients complete 1 course in the absence of unacceptable toxicity. Subsequent patients receive treatment on part 2.

Part 2: Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive monoclonal antibody SGN-30 IV over 2 hours, vinorelbine tartrate IV over 6-10 minutes, gemcitabine hydrochloride IV over 30 minutes, and pegylated doxorubicin hydrochloride liposome IV over 90 minutes on days 1 and 8.

Arm II (closed to accrual as of 12/4/07): Patients receive placebo IV over 2 hours, vinorelbine tartrate IV over 6-10 minutes, gemcitabine hydrochloride IV over 30 minutes, and pegylated doxorubicin hydrochloride liposome IV over 90 minutes on days 1 and 8.

Treatment in both arms repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

NOTE: Treatment with SGN-30/placebo was stopped on 4/12/2007 due to pulmonary toxicity.

After completion of study treatment, patients are followed up periodically for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented CD30-positive classical Hodgkin lymphoma according to the World Health Organization (WHO) classification of lymphoid malignancies that is recurrent or refractory after at least one prior therapy

  * Note: Patients with nodular lymphocyte predominant HL are not eligible; all other subtypes including nodular sclerosis, lymphocyte-depleted, lymphocyte rich, and mixed cellularity HL may be enrolled
  * Core needle biopsies are acceptable if they contain adequate tissue for primary diagnosis and immunophenotyping; bone marrow biopsies as the sole means of diagnosis are not acceptable, but they may be submitted in conjunction with nodal biopsies; fine needle aspirates are not acceptable; if the original diagnostic specimen is not available, specimens obtained at relapse may be submitted; if multiple specimens are available, please submit the most recent; failure to submit pathology specimens within 60 days of patient registration will be considered a major protocol violation
* Patients must have relapsed or refractory disease after at least one prior therapy, with at least a 3 week interval from the completion of the most recent chemotherapy or radiotherapy regimen; recovery to =< grade 1 from all toxicities related to the prior treatments is required; patients who have previously received a stem cell transplant are permitted to enroll on this study

  * Prior treatment with an anti-CD30 antibody, gemcitabine, vinorelbine, or pegylated liposomal doxorubicin is not permitted
* No uncontrolled angina, no myocardial infarction (MI) within 6 months of study entry, and no New York Heart Association (NYHA) class II or greater congestive heart failure (CHF)
* Baseline left ventricular ejection fraction (LVEF) by multi gated acquisition scan (MUGA) or echocardiogram (ECHO) must be >= 45%
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Measurable disease must be present on either physical examination or imaging studies; evaluable or non-measurable disease alone is not acceptable

  * Measurable disease is defined as any lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 10 mm
  * Non-measurable disease includes all other lesions, including small lesions (< 10 mm) and truly non-measurable lesions
  * Lesions that are considered non-measurable include the following:

    * Bone lesions (lesions, if present, should be noted)
    * Bone marrow involvement (if present, this should be noted)
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
* Pregnant or nursing women may not be enrolled; women of childbearing potential must have a negative serum or urine pregnancy test prior to registration; women and men of reproductive potential should agree to use an effective means of birth control
* Corrected diffusion capacity of carbon monoxide (DLCO) >= 50%
* Absolute neutrophil count (ANC) >= 1,200/uL
* Platelet count >= 100,000/uL
* Creatinine =< 2.0 mg/dL
* Bilirubin =< 2.0 mg/dL

  * Absent a history of Gilbert's disease
* Aspartate aminotransferase (AST) =< 2.0 x upper limits of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-04; Primary Completion 2008-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Blum, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2006 to December 2007 10 institutions recruited 30 participants to this trial.
Groups:
- Arm I (SGN-30, Chemotherapy): Participants receive one of the following regimens every cycle depending on history of prior stem cell transplant. Cycle is 21 days.
  No prior stem cell transplant:
  SGN-30: 12 mg/kg IV days 1 & 8, vinorelbine: 20 mg/m^2 IV days 1 & 8, gemcitabine: 1000 mg/m^2 IV days 1 & 8, pegylated doxorubicin HCl liposome: 15 mg IV days 1 & 8.
  Prior stem cell transplant SGN-30: 12 mg/kg IV days 1 & 8, vinorelbine: 15 mg/m^2 IV days 1 & 8, gemcitabine: 800 mg/m^2 IV days 1 & 8, pegylated doxorubicin HCl liposome: 10 mg IV days 1 & 8.
  monoclonal antibody SGN-30: Given IV
  vinorelbine tartrate: Given IV
  pegylated liposomal doxorubicin hydrochloride: Given IV
  gemcitabine hydrochloride: Given IV
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
- Arm II (Placebo, Chemotherapy): Participants receive one of the following regimens every cycle depending on history of prior stem cell transplant. Cycle is 21 days.
  No prior stem cell transplant:
  SGN-30: 12 mg/kg IV days 1 & 8, vinorelbine: 20 mg/m^2 IV days 1 & 8, gemcitabine: 1000 mg/m^2 IV days 1 & 8, pegylated doxorubicin HCl liposome: 15 mg IV days 1 & 8.
  Prior stem cell transplant SGN-30: 12 mg/kg IV days 1 & 8, vinorelbine: 15 mg/m^2 IV days 1 & 8, gemcitabine: 800 mg/m^2 IV days 1 & 8, pegylated doxorubicin HCl liposome: 10 mg IV days 1 & 8.
  placebo: Given IV
  vinorelbine tartrate: Given IV
  pegylated liposomal doxorubicin hydrochloride: Given IV
  gemcitabine hydrochloride: Given IV
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Period: Overall Study
Arm/Group | Arm I (SGN-30, Chemotherapy) | Arm II (Placebo, Chemotherapy)
Started | 23 | 7
Completed | 11 | 3
Not Completed | 12 | 4
Not completed — Adverse Event | 5 | 1
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Disease progression | 1 | 2
Not completed — Subsequent non-protocol therapy | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (SGN-30, Chemotherapy) | Arm II (Placebo, Chemotherapy) | Total
Number analyzed (Participants) | 23 | 7 | 30
Age, Continuous [Median (Full Range); unit: years] | 35 [19 to 78] | 38 [25 to 53] | 35 [19 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 18 | 5 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 18 | 6 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 7 | 30
Prior autologous transplant [Number; unit: participants]
  Yes | 8 | 3 | 11
  No | 15 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response (OR)
Description: The number of participants who respond (complete or partial) to treatment. Response was defined using the revised criteria for malignant lymphoma. Complete response (CR): complete disappearance of all detectable disease; partial response (PR): >= 50% reduction in sum of the product of diameters of indicator lesions.
Time Frame: Up to 10 years
Measure: Number; unit: participants
Arm/Group | Arm I (SGN-30, Chemotherapy) | Arm II (Placebo, Chemotherapy)
Number analyzed (Participants) | 23 | 7
participants | 15 | 4

2. Secondary Outcome: Event Free Survival (EFS)
Description: Event free survival is the time from trial entry until progression, death, or termination of treatment due to nonresponse. Patients who went on to receive a stem cell transplant (SCT) were not censored from the EFS survival at the time of transplant and were only considered failures at the time of relapse or death from any cause. The median EFS with 95% confidence interval (CI) was estimated using the Kaplan Meier method.
Time Frame: Up to 10 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (SGN-30, Chemotherapy) | Arm II (Placebo, Chemotherapy)
Number analyzed (Participants) | 23 | 7
months | 11.3 [4.7 to NA] — he upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 4.1 [1.8 to NA] — he upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

3. Secondary Outcome: Overall Survival (OS) At 1 Year
Description: Percentage of patients who were alive at 1 year. The 1-year survival rate was estimated using the Kaplan Meier method.
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (SGN-30, Chemotherapy) | Arm II (Placebo, Chemotherapy)
Number analyzed (Participants) | 23 | 7
percentage of participants | 86 [61 to 95] | 30 [13 to 72]

4. Other Pre Specified Outcome: Peak Serum Level of Monoclonal Antibody SGN-30
Description: Record the highest serum level of monoclonal antibody SGN-30 achieved.
Time Frame: Up to day 21 of course 6
Population: Data was only available on 10 participants from Arm 1. (No participants from Arm II were evaluable for this endpoint as they did not receive SGN-30 per protocol.)
Measure: Median (Full Range); unit: mg/ml
Arm/Group | Arm I (SGN-30, Chemotherapy)
Number analyzed (Participants) | 10
mg/ml | 339 [141 to 565]

5. Other Pre Specified Outcome: sCD30 Levels
Description: A 2-sided t-test with alpha = 0.05 will be used to compare sCD30 levels between responders (OR) and non-responders groups.
Time Frame: Up to day 21 of course 6
Population: Nine participants submitted pretreatment sCD30 samples.
Measure: Median (Full Range); unit: U/ml
Groups:
- Responders: Subset of patients who achieved an overall response, as describer in primary outcome measure 1.
- Non-responders: Subset of patients who did not achieve an overall response, as defined in primary outcome measure 1
Arm/Group | Responders | Non-responders
Number analyzed (Participants) | 4 | 5
U/ml | 174.2 [14.3 to 1992.0] | 76.5 [21 to 219.0]
Statistical Analysis 1: Comparison: Responders vs Non-responders; Test type: Superiority or Other; p = 0.06, Chi-squared

6. Other Pre Specified Outcome: Fc Gamma Receptor Polymorphisms
Description: Fisher's exact test with 2-sided alpha = 0.05 will be used to compare the response probabilities in patients with V/V (valine expression), V/F (heterozygous), and F/F (homozygous for phenylalanine) for each of Fc gamma RIIIa a
Time Frame: Baseline
Population: Fc gamma receptor polymorphisms were assessed in 28 participants.
Measure: Number; unit: participants
Arm/Group | Responders | Non-responders
Number analyzed (Participants) | 17 | 11
participants
  V/V | 0 | 0
  F/F | 10 | 6
  F/V | 7 | 5
Statistical Analysis 1: Comparison: Responders vs Non-responders; Test type: Superiority or Other; p = 1.0, Fisher Exact

ADVERSE EVENTS:
Groups:
- Arm II (Placebo, Chemotherapy): Participants receive one of the following regimens every cycle depending on history of prior stem cell transplant. Cycle is 21 days.
  No prior stem cell transplant:
  SGN-30: 12 mg/kg IV days 1 & 8, vinorelbine: 20 mg/m^2 IV days 1 & 8, gemcitabine: 1000 mg/m^2 IV days 1 & 8, pegylated doxorubicin HCl liposome: 15 mg IV days 1 & 8.
  Prior stem cell transplant SGN-30: 12 mg/kg IV days 1 & 8, vinorelbine: 15 mg/m^2 IV days 1 & 8, gemcitabine: 800 mg/m^2 IV days 1 & 8, pegylated doxorubicin HCl liposome: 10 mg IV days 1 & 8.
  placebo: Given IV
  vinorelbine tartrate: Given IV
  pegylated liposomal doxorubicin hydrochloride: Given IV
  gemcitabine hydrochloride: Given IV
  laboratory biomarker analysis: Correlative studies
  pharma
Arm/Group | Arm I (SGN-30, Chemotherapy) | Arm II (Placebo, Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 9/23 | 1/7
Other Adverse Events (participants affected / at risk) | 21/23 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (SGN-30, Chemotherapy) (N=23) | Arm II (Placebo, Chemotherapy) (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 6 (6) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0)
Fever (General disorders) | 4 (4) | 0 (0)
Visceral edema (General disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1)
Alkaline phosphatase increased (Investigations) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Laboratory test abnormal (Investigations) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 4 (4) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (5) | 1 (1)
Platelet count decreased (Investigations) | 4 (4) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Body odor (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (SGN-30, Chemotherapy) (N=23) | Arm II (Placebo, Chemotherapy) (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 15 (31) | 5 (8)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac pain (Cardiac disorders) | 1 (1) | 0 (0)
Edema (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (6) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 4 (5) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (16) | 4 (5)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Chest pain (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 3 (3) | 0 (0)
Edema limbs (General disorders) | 3 (6) | 2 (2)
Fatigue (General disorders) | 8 (13) | 6 (6)
Fever (General disorders) | 5 (6) | 0 (0)
Joint- Late RT Morbidity Scoring (General disorders) | 1 (2) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (3) | 0 (0)
Visceral edema (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Upper aerodigestive tract infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 9 (12) | 4 (6)
Alkaline phosphatase increased (Investigations) | 4 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 8 (12) | 3 (5)
Coagulopathy (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
INR increased (Investigations) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 10 (15) | 4 (7)
Lymphocyte count decreased (Investigations) | 7 (11) | 2 (4)
Neutrophil count decreased (Investigations) | 16 (21) | 6 (8)
Platelet count decreased (Investigations) | 16 (32) | 3 (7)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 3 (5) | 2 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 5 (9) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (5) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 8 (16) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 2 (6) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less